CLINICAL TRIAL: NCT04814589
Title: Bioequivalence of Ezetimibe Tablets in Healthy Subjects: A Single-dose and Two-period Crossover Study
Brief Title: Bioequivalence of Ezetimibe Tablets in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cao Yu (Other)
Responsible Party: Sponsor-Investigator, Cao Yu, Director, Head of Phase I clinical research center, Principal Investigator, Clinical Professor., The Affiliated Hospital of Qingdao University
Organization: The Affiliated Hospital of Qingdao University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: LC00-065
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Therapeutic Equivalency
MeSH Terms: interventions — Ezetimibe

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ezetimibe Tablets (Experimental): ezetimibe tablets test formulation at a single dose of 10 mg
  Interventions: Drug: ezetimibe tablets
- ezetimibe tablets(Ezetrol ®) (Active Comparator): ezetimibe tablets reference formulation at a single dose of 10 mg
  Interventions: Drug: ezetimibe tablets(Ezetrol ®)

INTERVENTIONS:
Drug: ezetimibe tablets — The subjects randomly received single oral administration of ezetimibe tablets 10 mg.
  Arms: ezetimibe Tablets
Drug: ezetimibe tablets(Ezetrol ®) — The subjects randomly received single oral administration of ezetimibe tablets 10 mg.
  Arms: ezetimibe tablets(Ezetrol ®)

SUMMARY:
According to the relevant provisions of bioequivalence test, ezetimibe Tablets (test preparation, T, 10mg / tablet) provided by China Resources Saike Pharmaceutical Co., Ltd. were compared with Ezetrol ® (reference preparation, R, 10mg / tablet) produced by MSD Pharma (Singapore) Pte. Ltd. to evaluate the bioequivalence of single dose in healthy subjects under fasting and fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects ≥18 years of age, with appropriate sex ratio;
* The body mass index is in the range of 19.0-26.0 kg/m2 (including the critical value). The weight of male is not less than 50.0 kg, and that of female is not less than 45.0 kg.
* The following examination show that the indicators are normal or abnormal without clinical significance. The examination including: Vital signs, physical examination, blood routine, blood biochemistry, urinalysis, pregnancy test for female, serological tests for hepatitis B virus, hepatitis C virus, human immunodeficiency virus (HIV), and syphilis virus, 12 lead ECG, breath test for alcohol, drug abuse test and Nicotine test.
* The subjects have no family planning within 3 months and could select contraceptive method.
* Before the study, all subjects have been informed of the study's purpose, protocal, benefits, and risks, and signed the informed consent voluntarily.

Exclusion Criteria:

* Alanine aminotransferase >1.0×ULN ,Aspartate aminotransferase >1.0×ULN or Total bilirubin >1.0×ULN.
* Subjects with allergic constitution.
* Being allergy to the study medications, smoking, alcohol abuse.
* Participation in another clinical trial within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-03-13 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 90 days
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC)0-t | 90 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-t
Area under the plasma concentration versus time curve (AUC)0-∞ | 90 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-∞

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 90 days
  Collection of adverse events
Incidence of abnormal blood pressure | 90 days
  Monitor both systolic and diastolic blood pressure
Incidence of abnormal temperature | 90 days
  Monitor the temperature

CONTACTS AND LOCATIONS:
Overall Officials: yu Cao, doctor, Principal Investigator — the study director of phase I clinical research center
Locations (1):
- Phase Ⅰ Clinical Research Center, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No